CLINICAL TRIAL: NCT00641667
Title: A Phase III Study of JNS020QD in Cancer Pain Patients - Evaluation of the Efficacy and Safety of JNS020QD Switched From Opioid Analgesics
Brief Title: An Efficacy and Safety Study of Fentanyl (JNS020QD) in Participants With Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014896; JNS020QD-JPN-C01
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Results first posted 2013-05-08 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-05

CONDITIONS: Pain; Cancer
Keywords: Pain; Cancer; Fentanyl; JNS020QD
MeSH Terms: conditions — Pain; Neoplasms | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fentanyl (Experimental)
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Fentanyl 1-day application transdermal patch releasing the drug at the rate of 12.5 microgram per hour (mcg/hr) to 100 mcg/hr applied once daily, and maintained for 2 days. Dose escalation or reduction is as per Investigator's discretion (maximum applied dose is 300 mcg/hr) up to Day 7 and then dose is fixed for next 3 days that is Day 10 (end of treatment period).
  Other Names: JNS020QD

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of fentanyl one-day transdermal patch (patch containing a drug that is put on the skin so the drug will enter the body through the skin) in participants switched from morphine preparations, oral oxycodone preparations, fentanyl citrate injection or fentanyl patch for cancer pain.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center (conducted in more than one center) and non-comparative study of fentanyl one-day transdermal patch. The study consists of 3 periods: Pre-treatment observation period (4-7 days), Treatment period (10 days) and Follow-up period (2 days). Treatment will be initiated at 12.5 microgram per hour (mcg/hr) and the initial dose of fentanyl will be determined based on the daily dose of the opioid analgesic taken by the participant before entering the study and will be maintained for 2 days to ensure safety of participants. Dose escalation or reduction will be as per the Investigator's discretion from Day 3 to Day 7 and thereafter dose will be again maintained from Day 7 to Day 9, ranging from 12.5 mcg/hr-100 mcg/hr and the maximum application dose will be 300 mcg/hr. The patch will be applied on areas including the chest, abdomen, upper arm or thigh and will be replaced daily for 10 days (a total of 9 applications; including the day of final patch removal). Efficacy will primarily be evaluated by visual analog scale (VAS) score. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants receiving any of the following drugs at a stable dose for at least 3 days (or 9 days in case of fentanyl patch) before the start of application of the study drug: Morphine preparations at less than or equal to 314 milligram per day (mg/day) as an oral morphine equivalent dose of less than or equal to 157 mg/day for suppository or less than or equal to 104 mg/day for injection, oral oxycodone preparations at less than or equal to 209 mg/day, fentanyl citrate injection at less than or equal to 2.0 mg/day, fentanyl patch less than or equal to 7.5 mg
* Participants assumed to use not more than 2 rescue doses (dose of a fast-acting opioid analgesic except fentanyl preparations used for lack of analgesic effect) daily for at least 3 days before the start of application of the study drug
* Participants showing a pain intensity of less than or equal to 34 millimeter (mm) on a 100-mm visual analog scale (VAS)
* Participants who have an established diagnosis of cancer and are notified of the disease
* Participants who can be hospitalized during the course of application of the study drug

Exclusion Criteria:

* Participants with impaired respiratory function due to chronic lung disease or others
* Participants with asthma (breathing disorder in which there is wheezing and difficulty in breathing or participants with bradyarrhythmia (slow, irregular heartbeats)
* Participants with following measurements indicative of hepatic or renal impairment during the pre-treatment observation period: Aspartate transaminase (AST) greater than 5 times the upper limit of reference range, Alanine transaminase (ALT) greater than 5 times the upper limit of reference range, serum creatinine greater than 3 times the upper limit of reference range
* Participants with any cerebral damage, such as brain tumor, accompanied by increased intracranial pressure, disturbance of consciousness, coma, or respiratory disturbance
* Participants with a history of hypersensitivity to fentanyl or other opioid analgesics

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Kitakyushu, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Fentanyl: Fentanyl 1-day application transdermal patch (patch containing a drug that was put on the skin so the drug entered the body through the skin) releasing the drug at the rate of 12.5 microgram per hour (mcg/hr) to 100 mcg/hr applied once daily, and maintained for 2 days. Dose escalation or reduction was as per Investigator's discretion (maximum applied dose was 300 mcg/hr) up to Day 7 and then dose was fixed for next 3 days that is Day 10 (end of treatment period).
Period: Overall Study
Arm/Group | Fentanyl
Started | 66
Completed | 60
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Worsening of underlying disease | 3

BASELINE CHARACTERISTICS:
Arm/Group | Fentanyl
Number analyzed (Participants) | 66
Age Continuous [Mean (Standard Deviation); unit: Years] | 63.80 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Pain Control
Description: Pain control was assessed based on change in Visual Analog Scale (VAS) and number of daily rescue doses during 3 days before completion of study drug from 3 days before start of study drug. For VAS score, a difference of less than or equal to +15 millimeter (mm) and for rescue doses, a difference of less than or equal to 1 was considered significant to achieve pain control. Pain Intensity VAS ranged from 0 mm (no pain) to 100 mm (severest pain conceivable) and rescue dose was defined as dose of fast-acting opioid analgesic (except fentanyl preparations) used for lack of analgesic effect.
Time Frame: Day 10 or early discontinuation (ED)
Population: Full Analysis Set (FAS) population included all participants who applied at least 1 study drug patch and had 1 VAS assessment performed after application of the study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 66
Percentage of Participants | 81.8 [70.4 to 90.2]

2. Secondary Outcome: Number of Participants With Response Based on Patient's Global Assessment Scale
Description: Participants were asked to assess their satisfaction with respect to the therapeutic efficacy (effectiveness) of the study drug on a 5-point scale ranging from 1 to 5, where 1 = extremely satisfied, 2 = satisfied, 3 = neither satisfied nor dissatisfied, 4 = dissatisfied and 5 = extremely dissatisfied.
Time Frame: Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10 or ED
Population: The FAS population included all participants who applied at least 1 study drug patch and had 1 VAS assessment performed after application of the study drug. 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Number; unit: Participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 66
Participants
  Day 1; Extremely satisfied (n=66) | 8
  Day 1; Satisfied (n=66) | 35
  Day 1; Neither satisfied nor dissatisfied (n=66) | 19
  Day 1; Dissatisfied (n=66) | 4
  Day 1; Extremely dissatisfied (n=66) | 0
  Day 2; Extremely satisfied (n=65) | 8
  Day 2; Satisfied (n=65) | 31
  Day 2; Neither satisfied nor dissatisfied (n=65) | 24
  Day 2; Dissatisfied (n=65) | 2
  Day 2; Extremely dissatisfied (n=65) | 0
  Day 3; Extremely satisfied (n=65) | 8
  Day 3; Satisfied (n=65) | 25
  Day 3; Neither satisfied nor dissatisfied (n=65) | 25
  Day 3; Dissatisfied (n=65) | 7
  Day 3; Extremely dissatisfied (n=65) | 0
  Day 4; Extremely satisfied (n=64) | 9
  Day 4; Satisfied (n=64) | 28
  Day 4; Neither satisfied nor dissatisfied (n=64) | 24
  Day 4; Dissatisfied (n=64) | 3
  Day 4; Extremely dissatisfied (n=64) | 0
  Day 5; Extremely satisfied (n=63) | 10
  Day 5; Satisfied (n=63) | 30
  Day 5; Neither satisfied nor dissatisfied (n=63) | 19
  Day 5; Dissatisfied (n=63) | 3
  Day 5; Extremely dissatisfied (n=63) | 1
  Day 6; Extremely satisfied (n=63) | 9
  Day 6; Satisfied (n=63) | 31
  Day 6; Neither satisfied nor dissatisfied (n=63) | 20
  Day 6; Dissatisfied (n=63) | 3
  Day 6; Extremely dissatisfied (n=63) | 0
  Day 7; Extremely satisfied (n=63) | 10
  Day 7; Satisfied (n=63) | 31
  Day 7; Neither satisfied nor dissatisfied (n=63) | 18
  Day 7; Dissatisfied (n=63) | 4
  Day 7; Extremely dissatisfied (n=63) | 0
  Day 8; Extremely satisfied (n=62) | 10
  Day 8; Satisfied (n=62) | 30
  Day 8; Neither satisfied nor dissatisfied (n=62) | 19
  Day 8; Dissatisfied (n=62) | 3
  Day 8; Extremely dissatisfied (n=62) | 0
  Day 9; Extremely satisfied (n=62) | 11
  Day 9; Satisfied (n=62) | 32
  Day 9; Neither satisfied nor dissatisfied (n=62) | 17
  Day 9; Dissatisfied (n=62) | 2
  Day 9; Extremely dissatisfied (n=62) | 0
  Day 10/ED; Extremely satisfied (n=66) | 10
  Day 10/ED; Satisfied (n=66) | 30
  Day 10/ED;Neither satisfied nor dissatisfied(n=66) | 20
  Day 10/ED; Dissatisfied (n=66) | 6
  Day 10/ED; Extremely dissatisfied (n=66) | 0

3. Secondary Outcome: Pain Intensity Visual Analog Scale (VAS) Score
Description: Participants were asked to assess their resting pain intensity (severity of pain) on a 100-mm VAS with the left edge (0 mm) defined as "no pain" and the right edge (100 mm) defined as "severest pain conceivable".
Time Frame: Day 1 (pre-application), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10 or ED
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Fentanyl
Number analyzed (Participants) | 66
mm
  Day 1 pre-application; (n=66) | 15.6 (11.77)
  Day 2; (n=65) | 16.1 (11.95)
  Day 3; (n=65) | 18.6 (15.84)
  Day 4; (n=64) | 15.1 (13.09)
  Day 5; (n=63) | 15.2 (14.31)
  Day 6; (n=63) | 15.3 (12.68)
  Day 7; (n=63) | 14.7 (13.47)
  Day 8; (n=62) | 14.9 (14.34)
  Day 9; (n=62) | 15.1 (13.38)
  Day 10 or ED; (n=66) | 15.5 (13.34)

4. Secondary Outcome: Number of Participants With Pain Intensity Assessed by Categorical Scale for Pain
Description: Participants were asked to assess their resting pain intensity (severity of pain) on a 4-point categorical scale ranging from 0 to 3 where 0 = no pain, 1 = mild pain, 2 = moderate pain and 3 = severe pain.
Time Frame: Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10 or ED
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 66
Participants
  Day 1; No pain (n=66) | 12
  Day 1; Mild pain (n=66) | 37
  Day 1; Moderate pain (n=66) | 17
  Day 1; Severe pain (n=66) | 0
  Day 2; No pain (n=65) | 10
  Day 2; Mild pain (n=65) | 34
  Day 2; Moderate pain (n=65) | 21
  Day 2; Severe pain (n=65) | 0
  Day 3; No pain (n=65) | 14
  Day 3; Mild pain (n=65) | 33
  Day 3; Moderate pain (n=65) | 15
  Day 3; Severe pain (n=65) | 3
  Day 4; No pain (n=64) | 16
  Day 4; Mild pain (n=64) | 34
  Day 4; Moderate pain (n=64) | 13
  Day 4; Severe pain (n=64) | 1
  Day 5; No pain (n=63) | 15
  Day 5; Mild pain (n=63) | 36
  Day 5; Moderate pain (n=63) | 12
  Day 5; Severe pain (n=63) | 0
  Day 6; No pain (n=63) | 16
  Day 6; Mild pain (n=63) | 38
  Day 6; Moderate pain (n=63) | 8
  Day 6; Severe pain (n=63) | 1
  Day 7; No pain (n=63) | 14
  Day 7; Mild pain (n=63) | 38
  Day 7; Moderate pain (n=63) | 11
  Day 7; Severe pain (n=63) | 0
  Day 8; No pain (n=62) | 13
  Day 8; Mild pain (n=62) | 38
  Day 8; Moderate pain (n=62) | 11
  Day 8; Severe pain (n=62) | 0
  Day 9; No pain (n=62) | 14
  Day 9; Mild pain (n=62) | 40
  Day 9; Moderate pain (n=62) | 7
  Day 9; Severe pain (n=62) | 1
  Day 10 or ED; No pain (n=66) | 15
  Day 10 or ED; Mild pain (n=66) | 40
  Day 10 or ED; Moderate pain(n=66) | 8
  Day 10 or ED; Severe pain(n=66) | 3

5. Secondary Outcome: Number of Participants With Total Duration of Pain Per Day
Description: The participants assessed total painful time in 1 day on a 5-point scale ranging from 0 to 4 where 0 = less than (<) 4 hours, 1 = greater than or equal to (>=) 4 hours to less than 8 hours, 2 = greater than or equal to 8 hours to less than 12 hours, 3 = greater than or equal to 12 hours and 4 = 24 hours (all day).
Time Frame: Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10 or ED
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 66
Participants
  Day 1; < 4 hours (n=66) | 44
  Day 1; >= 4 to < 8 hours (n=66) | 9
  Day 1; >= 8 to < 12 hours (n=66) | 6
  Day 1; >= 12 hours (n=66) | 0
  Day 1; 24 hours (n=66) | 7
  Day 2; < 4 hours (n=65) | 44
  Day 2; >= 4 to < 8 hours (n=65) | 9
  Day 2; >= 8 to < 12 hours (n=65) | 6
  Day 2; >= 12 hours (n=65) | 1
  Day 2; 24 hours (n=65) | 5
  Day 3; < 4 hours (n=65) | 41
  Day 3; >= 4 to < 8 hours (n=65) | 6
  Day 3; >= 8 to < 12 hours (n=65) | 9
  Day 3; >= 12 hours (n=65) | 3
  Day 3; 24 hours (n=65) | 6
  Day 4; < 4 hours (n=64) | 47
  Day 4; >= 4 to < 8 hours (n=64) | 8
  Day 4; >= 8 to < 12 hours (n=64) | 2
  Day 4; >= 12 hours (n=64) | 2
  Day 4; 24 hours (n=64) | 5
  Day 5; < 4 hours (n=63) | 45
  Day 5; >= 4 to < 8 hours (n=63) | 10
  Day 5; >= 8 to < 12 hours (n=63) | 2
  Day 5; >= 12 hours (n=63) | 1
  Day 5; 24 hours (n=63) | 5
  Day 6; < 4 hours (n=63) | 46
  Day 6; >= 4 to < 8 hours (n=63) | 6
  Day 6; >= 8 to < 12 hours (n=63) | 3
  Day 6; >= 12 hours (n=63) | 1
  Day 6; 24 hours (n=63) | 7
  Day 7; < 4 hours (n=63) | 44
  Day 7; >= 4 to < 8 hours (n=63) | 7
  Day 7; >= 8 to < 12 hours (n=63) | 4
  Day 7; >= 12 hours (n=63) | 1
  Day 7; 24 hours (n=63) | 7
  Day 8; < 4 hours (n=62) | 44
  Day 8; >= 4 to < 8 hours (n=62) | 6
  Day 8; >= 8 to < 12 hours (n=62) | 4
  Day 8; >= 12 hours (n=62) | 1
  Day 8; 24 hours (n=62) | 7
  Day 9; < 4 hours (n=62) | 47
  Day 9; >= 4 to < 8 hours (n=62) | 6
  Day 9; >= 8 to < 12 hours (n=62) | 3
  Day 9; >= 12 hours (n=62) | 1
  Day 9; 24 hours (n=62) | 5
  Day 10 or ED; < 4 hours (n=66) | 50
  Day 10 or ED; >=4 to < 8 hours (n=66) | 6
  Day 10 or ED; >=8 to <12 hours (n=66) | 3
  Day 10 or ED; >= 12 hours (n=66) | 2
  Day 10 or ED; 24 hours (n=66) | 5

6. Secondary Outcome: Mean Number of Rescue Doses
Description: Rescue dose was defined as the dose of a fast-acting opioid analgesic (except fentanyl preparations) given in case of breakthrough pain or lack of analgesic effect.
Time Frame: Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10 or ED
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Rescue Doses
Arm/Group | Fentanyl
Number analyzed (Participants) | 66
Rescue Doses
  Day 1; (n=66) | 0.2 (0.47)
  Day 2; (n=65) | 0.8 (1.06)
  Day 3; (n=65) | 0.7 (1.14)
  Day 4; (n=64) | 0.7 (1.04)
  Day 5; (n=63) | 0.7 (1.05)
  Day 6; (n=63) | 0.7 (1.10)
  Day 7; (n=63) | 0.8 (1.42)
  Day 8; (n=62) | 0.7 (1.14)
  Day 9; (n=62) | 0.8 (1.33)
  Day 10 or ED; (n=66) | 0.5 (0.83)

7. Secondary Outcome: Number of Participants With Response Based on Physician's Global Assessment Scale
Description: The treating physician assessed the therapeutic efficacy (effectiveness) of the study drug by 2-point scale of effective and ineffective. Number of participants with effective and ineffective therapeutic efficacy with respect to the study drug were reported.
Time Frame: Day 10 or ED
Population: The FAS population included all participants who applied at least 1 study drug patch and had 1 VAS assessment performed after application of the study drug.
Measure: Number; unit: Participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 66
Participants
  Effective | 63
  Ineffective | 3

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to 7 days after the completion or discontinuation of last study treatment
Arm/Group | Fentanyl
Serious Adverse Events (participants affected / at risk) | 6/66
Other Adverse Events (participants affected / at risk) | 56/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl (N=66)
Pneumonia (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl (N=66)
Nasopharyngitis (Infections and infestations) | 4
Insomnia (Psychiatric disorders) | 5
Dizziness (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 36
Constipation (Gastrointestinal disorders) | 34
Diarrhoea (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 25
Vomiting (Gastrointestinal disorders) | 23
Erythema (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 6
Application site erythema (General disorders) | 4
Application site pruritus (General disorders) | 7
Pyrexia (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on PI is that the Sponsor can review results communications prior to public release and can embargo communications regarding results for a period as the Sponsor requires.